CLINICAL TRIAL: NCT07327879
Title: Comparative Efficacy and Dose-Response of Intrathecal Dexmedetomidine in Attenuating Post-Spinal Shivering: Double-Blinded Randomized Controlled Trial
Brief Title: Comparative Dose-Response of Intrathecal Dexmedetomidine for Post-Spinal Shivering
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC. 2.12.2025
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Post-Spinal Shivering
Keywords: Intrathecal Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group P (Placebo Comparator): Patients in this group will receive the standard spinal anesthetic consisting of hyperbaric bupivacaine 0.5% (15 mg) combined with an equivalent volume of normal saline (0.9% NaCl), containing no active dexmedetomidine. The total intrathecal injection volume will be standardized to 3.5 mL across all groups by adjusting the volume of saline added.
  Interventions: Drug: Group P (Placebo Control Group)
- Group D2.5 (Experimental): Patients in this group will receive the standard spinal anesthetic (15 mg hyperbaric bupivacaine 0.5%) supplemented with a low dose of 2.5 µg of dexmedetomidine. Normal saline will be added to achieve the standardized total intrathecal volume of 3.5 mL.
  Interventions: Drug: Group D2.5 (Low-Dose Dexmedetomidine Group)
- Group D5 (Experimental): Patients in this group will receive the standard spinal anesthetic combined with a moderate dose of 5 µg of dexmedetomidine. The total volume will be adjusted to 3.5 mL with normal saline.
  Interventions: Drug: Group D5 (Moderate-Dose Dexmedetomidine Group)
- Group D10 (Experimental): Patients in this group will receive the standard spinal anesthetic supplemented with a higher dose of 10 µg of dexmedetomidine, with normal saline used to standardize the total volume to 3.5 mL.
  Interventions: Drug: Group D10 (Higher-Dose Dexmedetomidine Group)

INTERVENTIONS:
Drug: Group P (Placebo Control Group) — Patients in this group will receive the standard spinal anesthetic consisting of hyperbaric bupivacaine 0.5% (15 mg) combined with an equivalent volume of normal saline (0.9% NaCl), containing no active dexmedetomidine. The total intrathecal injection volume will be standardized to 3.5 mL across all groups by adjusting the volume of saline added. This group serves as the control to establish the baseline incidence and characteristics of post-spinal shivering and block dynamics without the intervention of the α2-adrenergic agonist.
  Arms: Group P
Drug: Group D2.5 (Low-Dose Dexmedetomidine Group) — Patients in this group will receive the standard spinal anesthetic (15 mg hyperbaric bupivacaine 0.5%) supplemented with a low dose of 2.5 µg of dexmedetomidine. Normal saline will be added to achieve the standardized total intrathecal volume of 3.5 mL.
  Arms: Group D2.5
Drug: Group D5 (Moderate-Dose Dexmedetomidine Group) — Patients in this group will receive the standard spinal anesthetic combined with a moderate dose of 5 µg of dexmedetomidine. The total volume will be adjusted to 3.5 mL with normal saline.
  Arms: Group D5
Drug: Group D10 (Higher-Dose Dexmedetomidine Group) — Patients in this group will receive the standard spinal anesthetic supplemented with a higher dose of 10 µg of dexmedetomidine, with normal saline used to standardize the total volume to 3.5 mL.
  Arms: Group D10

SUMMARY:
Dexmedetomidine, a highly selective α2-adrenergic agonist, when used intrathecally as an adjuvant to local anesthetics, prolongs sensory/motor block and may blunt thermoregulatory shivering mechanisms. Several randomized controlled trials and meta-analyses have demonstrated decreased shivering incidence with intrathecal dexmedetomidine, but reported doses vary (commonly 2.5, 5, and 10 µg, and in some trials up to 15-20 µg), and the balance between efficacy and adverse effects (sedation, bradycardia, and hypotension) is not fully established. Hence, a head-to-head randomized comparison of several low-to-moderate intrathecal doses is warranted.

Objective: to compare the safety and efficacy of three intrathecal dexmedetomidine doses (2.5 µg, 5 µg, 10 µg) versus placebo for the prevention of post-spinal shivering.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-75 years)
* Scheduled for ureteric stone removal surgery
* ASA(American Society of Anesthesiologists) physical status I, II, or III
* Able to provide informed consent

Exclusion Criteria:

* Known allergy to dexmedetomidine, bupivacaine, or other study medications
* Preexisting bradycardia (heart rate <50 beats per minute)
* Second- or third-degree atrioventricular (AV) block without a pacemaker
* Severe hepatic dysfunction
* Uncontrolled hypotension
* Pregnancy
* Chronic use of α₂-agonists or antagonists (e.g., clonidine, tizanidine)
* Infection at the planned spinal puncture site
* Coagulopathy or bleeding disorder
* Inability to rate or communicate shivering (e.g., language barrier, cognitive impairment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically significant shivering | Throughout the intraoperative period until 60 minutes post-spinal.
  Incidence of clinically significant shivering within 60 minutes after spinal injection, defined as Crossley and Mahajan shivering scale grade ≥2 (scale 0-4)The highest intensity of shivering experienced by the patient, scored on the 0-4 scale. The Crossley and Mahajan shivering scale is a clinically validated, four-grade ordinal scale (0-4) used to objectively quantify the severity of post-anesthetic shivering. It is defined as follows: Grade 0 signifies no shivering; Grade 1 indicates mild, intermittent fasciculations of the face, neck, or chest; Grade 2 represents visible, intermittent shivering involving more than one muscle group; Grade 3 denotes generalized, continuous shivering of the whole body; and Grade 4 describes gross, bed-shaking tremors that interfere with monitoring or procedure. Grade ≥2 is typically considered clinically significant and often triggers therapeutic intervention. The scale is assessed through direct visual observation of the patient by trained personnel.

SECONDARY OUTCOMES:
Time to first shivering episode | Intraoperative period, up to 60 minutes post-spinal.
  The duration from the completion of the spinal injection to the onset of the first observable shivering (any grade).
Requirement of rescue anti-shivering drug | Intraoperative period, as needed.
  the number of patients required pharmacologic intervention (meperidine or tramadol) to treat severe shivering.
Dose of rescue anti-shivering drug | Intraoperative period, as needed.
  The total amount of pharmacologic intervention (meperidine or tramadol) to treat severe shivering.
Sedation level | Postoperative 24 hour
  The Ramsey Sedation Scale (RSS) is a simple, widely used six-level clinical tool (scores 1-6) for assessing a patient's level of sedation and responsiveness. It is scored as follows: 1 - Patient is anxious, agitated, or restless; 2 - Patient is cooperative, oriented, and tranquil; 3 - Patient responds only to commands; 4 - Patient exhibits a brisk response to a light glabellar tap or loud auditory stimulus; 5 - Patient exhibits a sluggish response to such a stimulus; and 6 - Patient exhibits no response to stimulus.
Patient satisfaction | Postoperatively (e.g., prior to discharge from PACU).
  The patient's overall satisfaction with the anesthesia experience.Using a Likert scale (e.g., 1-5 or 1-10) or a standardized satisfaction questionnaire.
Time to first analgesic request | 24 hours Postoperatively.
  The duration from the end of surgery until the patient first requires supplemental pain medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP